CLINICAL TRIAL: NCT02972086
Title: Improving Behavioral Health Care for Children With ADHD: Integration of Family Peer Advocates to Deliver Behavioral Parent Training in Pediatric Care Settings
Brief Title: Improving Behavioral Health Care for Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-01291
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent (Experimental): Parent of a child who is a patient at the NYU Bellevue Attention Deficit Hyperactivity Disorder (ADHD) Clinic
  Interventions: Behavioral: Behavioral Parent Training (BPT)

INTERVENTIONS:
Behavioral: Behavioral Parent Training (BPT) — A specific intervention modality that has been shown to improve key functional outcomes in youth with ADHD.

SUMMARY:
The purpose of this study is development of the Integrative Pediatric FPA ADHD Care (IPFAC) Model. The IPFAC is intended to increase access to evidence-based behavioral parent training (BPT) for school-age children diagnosed with attention-deficit/hyperactivity disorder(ADHD) who are diagnosed with ADHD and served in the ADHD Clinic at NYU Bellevue's Department of Developmental and Behavioral Pediatrics.

DETAILED DESCRIPTION:
The specific aims of this study are to: 1) Develop the IPFAC model (Phase I); 2) Assess and determine facilitators and barriers to fidelity, assess feasibility of data acquisition, determine preliminary efficacy, and refine the IPFAC model through a small-scale implementation study and Plan-Do-Study-Act methods (Phase II), and, 3) Evaluate the revised IPFAC model in a small-scale study using state-of-the-art single-case study design methods/analyses to test "treatment mechanisms" in a sample of newly diagnosed youth with ADHD (Phase III) and finalize the IPFAC procedural manual.

ELIGIBILITY:
Inclusion Criteria:

* being a parent of a child who is a patient at the NYU Bellevue ADHD Clinic
* being an adult over the age of 18
* having a child who obtained a diagnosis of ADHD (any subtype) within the previous 3 months (ie.., newly diagnosed) through the NYU Bellevue ADHD Clinic
* parent must speak English and/or Spanish.

The second study participant is the child. Study inclusion criteria for children include:

* child is a patient at the NYU Bellevue ADHD Clinic
* child is between the age of 6-11
* participating child must have obtained a diagnosis of ADHD (any subtype) within the previous 3 months (i.e., newly diagnosed) through the NYU Bellevue ADHD Clinic,
* child must speak English and/or Spanish.

Exclusion Criteria:

* parent presenting with severe mental health illness (e.g., schizophrenia; bipolar disorder) that would warrant immediate services.
* child with primary diagnosis/presenting issues of severe mental illness (e.g., schizophrenia; bipolar disorder) that would warrant primary services other than what is offered through the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01-07 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Attendance at BPT sessions | 16 Weeks
  Family Practice Associates (FPAs) will provide information on the extent to which the family attended scheduled BPT sessions.
Parenting Behavior | 16 Weeks
  The Alabama Parenting Questionnaire- Short Form (APQ-SF) is a well-validated 9-item measure of parenting style. Items are rated by the parent scored based on frequency of parenting behavior from Never (1), Almost Never (2), Sometimes (3), Often (4), Always (5). APQ-SF items are based around the three main structures: positive parenting, inconsistent discipline and poor supervision.
ADHD and oppositional behavior will be measured by the IOWA Connors Rating Scale (IOWA-CRS) | 16 Weeks
  The IOWA-CRS (Waschbusch & Willoughby, 2008) is a widely used brief measure of attention-deficit/hyperactivity disorder and oppositional-defiant behavior in children completed by parents. The IOWA-CRS consists of 10 items evaluated using a four-point Likert scale with the following anchors: not at all (0); just a little (1); pretty much (2); and very much (3).
Parental Depressive Symptoms using Beck Depression Inventory-II | 16 Weeks
  a 21-item self-report measure used to assess maternal depressive symptoms. Mothers were instructed to indicate which of four statements best described how they felt over the preceding two week period. The BDI is scored from one to four, with higher scores on the BDI indicating a greater degree of depression. A total score on the BDI, which is a sum of the 21-item measure, will be used in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hopkins, MD, Principal Investigator — NYU Langone Pediatric Department
Locations (1):
- New York University School of Medicine, New York, New York, United States